CLINICAL TRIAL: NCT04814043
Title: Systemic PD-1 Antibody (Sintilimab) and Lenvatinib Plus Transarterial Chemoembolization and FOLFOX-based Chemotherapy Infusion for Potential Resectable HCC: a Single-arm, Phase 2 Clinical Trial
Brief Title: PD-1 Antibody and Lenvatinib Plus TACE-HAIC for Potential Resectable HCC: a Single-arm, Phase 2 Clinical Trial
Acronym: PLATIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-411
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors; lenvatinib

STUDY DESIGN:
Intervention Model Description: systemic PD-1 antibody and lenvatinib plus TACE-HAIC for potential resectable HCC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody and lenvatinib plus TACE-HAIC (Experimental): systemic PD-1 antibody (Sintilimab) and lenvatinib plus transarterial chemobolization and FOLFOX-based chemotherapy infusion
  Interventions: Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: PD-1 inhibitor — systemic PD-1 antibody (Sintilimab) and lenvatinib plus transarterial chemobolization and FOLFOX-based chemotherapy infusion
  Other Names: lenvatinib; TACE-HAIC

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most commonly malignant tumors around the world. Hepatic resection or liver transplantation is the radical method to cure the disease. However, less than 20% of newly diagnosed patients can undergo radical resection. Our latest study showed that 48% potentially resectable HCC received hepatectomy after transarterial chemoembolization plus FOLFOX-based chemotherapy infusion (TACE-HAIC) treatment. Recently, several clinical trials (LEAP-002) showed that PD-1 antibody and Lenvatinib had an ORR of 36% for advanced patients. The combination of TACE-HAIC with PD-1 antibody and lenvatinib, theoretically can significantly decrease the tumor burden and increase the hepatectomy rate. However, this hasn't been verified in clinical application. To identify a more effective and safety way for treating potentially resectable HCC patients, this study is designed to investigate TACE-HAIC plus PD-1 antibody and Lenvatinib will increase the resection rate for those patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as potentially resectable with consensus by the panel of liver surgeons
* stage BCLC A/B/C, without extra-hepatic involvement
* No previous anti-HCC treatment
* Eastern Co-operative Group performance status 2 or less
* Liver function: Child's A or B (score < 7)

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy

  * underlying serve cardiac or renal diseases Known or suspected allergy to the investigational agent or any agent given in association with this trial
  * Patients ineligible for hepatic artery embolization, or PD-1 antibody

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
conversion rate to resection | 12 month
  The conversion rate to resection among all the enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Yuan, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No